CLINICAL TRIAL: NCT00816608
Title: Study of MAXimum Weight in Lifetime on Glucose Homeostasis (MAXWEL)
Brief Title: The Effect of Maximum Body Weight in Lifetime on the Development of Type 2 Diabetes
Acronym: MAXWEL
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Other Study IDs: MAXWEL 09
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes; Prediabetes
Keywords: diabetes; prediabetes; impaired fasting glucose (IFG); impaired glucose tolerance (IGT); body weight
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Glucose Intolerance; Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- type 2 diabetes

SUMMARY:
Hypothesis : The maximum body weight in lifetime is associated with the onset of development of type 2 diabetes.

DETAILED DESCRIPTION:
Obesity is well recognized risk factor for type 2 diabetes. Recent studies reported that weight change, especially severe weight gain was associated with an increased risk of type 2 diabetes. The aim of this study is to investigate whether the maximum body weight of lifetime is associated with the early onset of type 2 diabetes or an increased risk of type 2 diabetes in Korean.

ELIGIBILITY:
Inclusion Criteria:

* Korean with type 2 diabetes
* Korean with confirmed IFG or IGT
* Korean with NGT

Exclusion Criteria:

* Malignancy except thyroid cancer
* Active tuberculosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean with type 2 diabetes Korean with confirmed IFG or IGT Korean with NGT
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2006-08; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The development of diabetes | Five years

SECONDARY OUTCOMES:
DM complication | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Bundang-gu, South Korea